CLINICAL TRIAL: NCT00835562
Title: Effect of Osteosynthesis, Primary Hemi-arthroplasty, and Non-surgical Management for Displaced Four-part Fractures of the Proximal Humerus in Elderly: a Multi-centre, Randomised Clinical Trial
Brief Title: Effect of Osteosynthesis, Primary Hemi-arthroplasty, and Non-surgical Management for Fractures of the Proximal Humerus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Zealand University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stig Brorson, MD PhD, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shoulderfractures.RCT; H-C-2008-065
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Proximal Humeral Fractures
Keywords: Shoulder fractures; Proximal humeral fractures; Randomised clinical trial; elderly; Displaced four-part fractures of the proximal humerus
MeSH Terms: conditions — Shoulder Fractures | interventions — Fracture Fixation, Internal; Hemiarthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Osteosynthesis (Experimental)
  Interventions: Procedure: Osteosynthesis
- Non-surgical (Experimental)
  Interventions: Procedure: Non-surgical management
- Hemiarthroplasty (Experimental)
  Interventions: Procedure: Hemiarthroplasty

INTERVENTIONS:
Procedure: Non-surgical management — Non-surgical management (physiotherapy and self-training)
  Arms: Non-surgical
Procedure: Osteosynthesis — Osteosynthesis with angle-stable plate followed by physiotherapy and self-training
  Arms: Osteosynthesis
Procedure: Hemiarthroplasty — Primary modular hemiarthroplasty followed by physiotherapy and self-training
  Arms: Hemiarthroplasty

SUMMARY:
Displaced four-part fractures are among the most severe injuries of the proximal humerus. The optimal treatment is disputed and published data are inadequate for evidence-based decision making.

The investigators aim to: 1) compare the effect of angle-stable plate osteosynthesis and non-surgical management, 2) compare the effect of primary hemiarthroplasty with both osteosynthesis and non-surgical management, 3) study prognostic differences between 'valgus impacted' and 'classical' four-part fracture patterns.

The investigators will conduct a randomised, multi-centre, clinical trial including patients from ten national shoulder units within a two year period. Patients will be randomised to non-surgical treatment, hemiarthroplasty or angle-stable plate osteosynthesis. All patients will receive a standardised three-month rehabilitation program of supervised physiotherapy. Patients will be followed at least one year and will be assessed blindly according to a standardised evaluation protocol including Constant Disability Scale, Oxford Shoulder Score, and Short Form-36.

ELIGIBILITY:
Inclusion Criteria:

* Displaced four-part fracture of the proximal humerus
* Mentally alert
* Physically fit for surgery and rehabilitation (ASA-group 1-3)
* Informed written consent
* Operation can be conducted within 2 weeks of injury

Exclusion Criteria:

* Fracture-dislocations
* Head-splitting fractures
* Previous shoulder surgery on injured side
* Chronic shoulder pain
* Abuse problems
* Patients unable to understand instructions in Danish

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Constant Disability Scale | 3 years

SECONDARY OUTCOMES:
Oxford Shoulder Score, Short Form-36 | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev University Hospital, Department Orthopaedic Surgery, Herlev, Denmark, Denmark

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196